CLINICAL TRIAL: NCT02272439
Title: Endocrine Disrupting Chemicals: Potential Effects on Male and Female Reproductive Health in Saskatchewan.
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Angela Baerwald, Assistant Professor, University of Saskatchewan
Other Study IDs: EDC-ARB-002
Record Dates: First submitted 2013-04-11; First posted 2014-10-23 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Unexplained Infertility; Polycystic Ovarian Syndrome; Male Infertility
Keywords: Bisphenol A; phthalates; infertility; human
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — Blood, Follicular Fluid and Seminal Plasma Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Unexplained (male): Men of couples with a diagnosis of Unexplained infertility (n=15)
- Unexplained (female): Women of couples with a diagnosis of Unexplained infertility (n=15)
- male factor (male): Men of couples with a diagnosis of male factor infertility (n=15)
- male factor (female/control): Women of couples with a diagnosis of male factor infertility (n=15)
- PCOS (female): Women of couples with a diagnosis of Polycystic Ovarian Syndrome-related infertility (n=15)
- PCOS (male/control): Men of couples with a diagnosis of Polycystic Ovarian Syndrome-related infertility (n=15)
- healthy volunteer (male/control): Men with a history of no reproductive dysfunction and proven fertility (n=15)
- healthy volunteer (female/control): Women with a history of no reproductive dysfunction and proven fertility (n=15)

SUMMARY:
The overall objective of this study is to determine whether serum BPA and/or phthalate concentrations differ in fertile versus infertile men and women in Saskatchewan. The investigators will test the following hypothesis:

1. Serum BPA and/or phthalate concentrations will be greater in women with unexplained infertility or PCOS compared to a control group
2. Serum BPA and/or phthalate concentrations will be greater in men with male factor infertility compared to a control group

DETAILED DESCRIPTION:
Study Sample:

Couples undergoing in vitro fertilization (IVF) and/or Intracytoplasmic Sperm Injection (ICSI) for assisted reproduction at ARTUS as well as healthy male and female volunteers 18-43 years of age will be asked to participate. In order for infertility patients to be eligible, both the male and female partners must agree to participate. Couples with a combination of both male and female factor infertility will not be eligible to participate. Couples undergoing infertility treatment for the following reasons will be evaluated:

* unexplained infertility (n=15 men, n=15 women)
* PCOS (n=15 men, n=15 women)
* Male factor infertility (n=15 men, n=15 women)

Couples with male factor infertility will serve as controls for the female comparisons (i.e., follicular fluid analyses), and couples with PCOS will serve as controls for the male comparisons (i.e., seminal plasma analyses).

Additional participants will be assigned to the following control groups (for blood sample analyses):

-Healthy volunteers with no history or current diagnosis of reproductive dysfunction (n=15 men, n=15 women)

Participant Recruitment:

Infertile couples will be recruited from the clinical practices of Drs. Allison Case and Adrian Gamelin at the Assisted Reproductive Technologies Centre at the University of Saskatchewan (ARTUS). Posters for recruiting ARTUS patients will also be placed in the waiting room and examining rooms in the Dept of OB/GYN, Division of REI. Healthy male and female volunteers will be recruited from advertisements on the PAWS website at the University of Saskatchewan and Health E-News newsletters in the Saskatoon Health Region.

Pre-Study Visit:

Eligible participants will be asked to visit the ARTUS Centre for a pre-study appointment. At this appointment, study procedures will be discussed with participants and consent will be obtained.

Study Visits:

Blood and follicular fluid samples will be obtained from female partners of infertile couples. Blood and seminal plasma samples will be obtained from male partners of infertile couples. Only blood samples will be collected from healthy men and women. All samples will be collected in both fertile and infertile couples over a 2 week time interval.

A. Infertile couples:

Infertile couples participating in this study will undergo fertility treatment as per the normal standard of care. In other words, the fertility medications, ultrasound assessments, blood work during treatment, oocyte retrieval, semen collection, laboratory procedures and embryo transfer procedures will not be affected by participating in this study.

Both the male and female partner will be asked to provide 1 extra blood sample (approximately 7 mL or 1 teaspoon of blood) on each of the following regularly-scheduled appointments:

1. First ultrasound visit (approximately day 1 of FSH therapy)
2. Day of egg retrieval
3. Day of embryo transfer

Women normally undergo regular blood draws during their IVF treatment; therefore, one additional tube will be drawn for research purposes at the regularly-scheduled blood draw appointments. Men do not normally provide a blood sample during IVF treatment, but will be asked to do so in this study. Blood draws will be performed by phlebotomists (staff that specialize in drawing blood) at Royal University Hospital, physicians, nurses and/or researchers with training in phlebotomy. The blood samples will be processed to remove the cells, and the serum will be frozen for 12-24 months until the completion of the study.

The follicles in the woman's ovaries will be drained and the eggs will be retrieved from the follicular fluid, as per the standard of care. After the eggs are collected, the follicular fluid is normally thrown away. In this study, we will collect the fluid from the follicles on each ovary after the eggs are retrieved. The follicular fluid will be frozen for 12-24 months until study completion.

A semen sample will be provided by the man on the day of the oocyte retrieval procedure, as per standard of care. The semen sample is processed by allowing the semen to pass through a column to separate the most motile sperm (moving very quickly) from the less motile and non-motile sperm. The seminal plasma is the fluid portion of the semen that remains after the most motile sperm have been obtained. The seminal plasma is normally thrown away after the motile sperm are obtained. In this study, we will collect the seminal plasma and freeze it for 12-24 months until the study is completed.

B. Healthy Volunteers:

Healthy volunteers will be asked to provide 1 blood sample (approximately 7 mL or 1 teaspoon of blood) on 3 separate days. Blood draws will be performed by physicians, nurses and/or researchers with training in phlebotomy (i.e., drawing blood). Appointments for blood draws will be made approximately 4-7 days apart.

At the completion of the study all of the frozen blood, follicular fluid, and seminal plasma samples will be transported to the Toxicology Center at the University of Saskatchewan. The levels of exposure to BPA and phthalates will be evaluated. The samples will be destroyed upon completion of the study. The expected duration of study participation is approximately 13-20 days (in accordance with standard fertility therapy) for fertility patients and 3 days for healthy volunteers. All samples will be obtained over a 2 week time period.

Statistical Analysis

Include a summary of the primary and secondary end-points/outcomes, the planned sample size (with justification) and planned statistical and interim analyses.

Study Endpoints:

Exposure to phthalates will be determined by quantifying concentrations of 5 different pthalates. Concentrations of Bisphenol A (BPA), di-2-ethylhexyl phthalate (DEHP), di-n-octyl phthalate (DNOP), di-n-butyl phthalate (DNBP), n-butyl benzyl phthalate (BBP), diethyl phthalate (DEP), diisononyl phthalate (DINP) and diisodecyl phthalate (DIDP) will be quantified in the blood cells, blood plasma, and follicular fluid (individual and pooled samples) by use of liquid chromatography and tandem mass spectrometry methods already developed in our laboratory. Analyses will be conducted by use of an Agilent 1200 series High Performance Liquid Chromatography (HPLC) system interfaced to an ABI SCIEX 3200 triple quadrapole mass spectrometer system or to a QToF II quadrapole time of flight mass spectrometer (Micromass, Beverly MD). Toxicant concentrations will be the dependent variables. Reproductive status (i.e, unexplained infertility, PCOS, male factor infertility, controls) will be the independent variable. Concentrations of BPA and phthalates in blood cells, blood plasma, seminal plasma and pooled follicular fluid will be compared between study groups using multivariate Analyses of Variance (ANOVA).

n=15 per group is appropriate for conducting this pilot study.

Potential Significance/Justification:

Greater knowledge about the possible effects of BPA and phthalates on reproductive function may increase our understanding of the causes of infertility, assist in preventing reproductive disease, and optimize reproductive health, which will thereby improve patient care. We believe that the results of our study, whether positive or negative, will be of interest to the general public, health professionals and scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-43 years
* Couples undergoing IVF for:

Unexplained infertility Male factor infertility Polycystic Ovary(PCOS)

-Both male and female partners must agree to participate

Exclusion Criteria:

* Age: <18 and >43 years
* Couples with both male and female factor infertility
* Only female or male partner agrees to participate

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile couples with unexplained infertility, male factor infertility and PCOS Healthy volunteers with history of fertility
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Exposure to BPA | March 2012 to September 2013 (up to 2 years)
  Concentrations of Bisphenol A (BPA), di-2-ethylhexyl phthalate (DEHP), di-n-octyl phthalate (DNOP), di-n-butyl phthalate (DNBP), n-butyl benzyl phthalate (BBP), diethyl phthalate (DEP), diisononyl phthalate (DINP) and diisodecyl phthalate (DIDP) will be quantified in the blood cells, blood plasma, and follicular fluid (individual and pooled samples) by use of liquid chromatography and tandem mass spectrometry methods and will be compared between study groups using multivariate Analyses of Variance (ANOVA).

SECONDARY OUTCOMES:
Exposure to Phthalates | March 2012 to Sep. 2013 (up to 2 years)
  Exposure to phthalates will be determined by quantifying concentrations of 5 different pthalates. Concentrations of BPA and phthalates in blood cells, blood plasma, seminal plasma and pooled follicular fluid will be compared between study groups using multivariate Analyses of Variance (ANOVA).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Baerwald, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Obstretrics, Gynecology and Reproductive Science, RUH, Saskatoon, Saskatchewan, Canada